CLINICAL TRIAL: NCT03443310
Title: A Pilot Study of Bedside Ultrasound by Anesthesiologists for Screening Deep Venous Thrombosis in High Risk Patients Following Hip Fracture and Major Joint Arthroplasty
Brief Title: Bedside Ultrasound by Anesthesiologists for Screening Deep Venous Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11-0384-A
Record Dates: First submitted 2013-02-11; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: DVT
Keywords: DVT; TKA; THA; Hip Fracture; High risk; Ultrasound; U/S
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Patients who have symptomatic DVT undergo diagnostic venous duplex examination.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound assessment of DVT (Other): DVT ultrasound vs Clinical assessment in high-risk patients following hip fracture and major arthroplasty before the patients become symptomatic.
  Interventions: Procedure: Ultrasound assessment of DVT

INTERVENTIONS:
Procedure: Ultrasound assessment of DVT — Using Ultrasound in assessing DVT in high-risk patients following hip fracture and major arthroplasty before the patients become symptomatic.

SUMMARY:
The study is designed as a prospective comparative study. All patients will receive prophylactic anticoagulation according to routine hospital protocol after surgery. A bedside ultrasound examination will be performed by a trained anesthesiologist prior to the surgery and then daily beginning on postoperative day 2 until patient discharge.

DETAILED DESCRIPTION:
Recent studies conducted at the emergency department evaluated the usefulness of an abbreviated bedside compression ultrasound test for diagnosis of Deep Venous Thrombosis (DVT) in the proximal region. This abbreviated ultrasound test conducted in the groin and popliteal regions to assess the compressibility of the femoral and popliteal veins required as little as 3.5 min to complete 15 and can be easily mastered by residents with minimum training. These studies showed a promising sensitivity ranging from 70% to 100% and a specificity ranging from 75.9% to 99.6%.

Anesthesiologists are now well-trained in performing ultrasound scans as they perform ultrasound-guided peripheral nerve blocks routinely. Scanning for significant proximal DVT could potentially be anesthesiologists' extended role as they follow up patients who underwent orthopedic surgeries for postoperative pain control as part of the acute pain service.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* 18-85 years of age, inclusive
* 50-110 kg, inclusive
* 150 cm of height or greater
* Patients who are scheduled to have surgical repair of the fractured hip and those who will have unilateral or bilateral, primary or revision, hip or knee arthroplasty.

Exclusion Criteria:

* The presence of indwelling femoral vascular catheter or dialysis vascular shunts in the operative leg
* An above-knee amputation
* The inability to access all two landmarks (femoral and popliteal veins) for two-point ultrasonography because of the presence of a cast, external fixation apparatus, or other obstacles

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The accuracy of a positive bedside ultrasound scan | post operative day 2
  To evaluate the accuracy of a positive bedside ultrasound scan as compared to clinical assessment for the detection of an occluding DVT.

SECONDARY OUTCOMES:
The degree of technical difficulty | from start to of bedside compression test up to 1 hour
  The degree of technical difficulty in visualizing relevant veins and in determining whether a clot is present. That is, the incidence of uninterpreted test data in patients with a swollen thigh/leg after major hip or knee surgery. The degree of technical difficulty will be recorded especially in patients with a high body mass index (BMI).

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hopspital, Toronto, Ontario, Canada